CLINICAL TRIAL: NCT03258918
Title: A Mixed Methods Pilot Study of a Low-Carbohydrate Diabetes Prevention Program Among Individuals With Prediabetes
Brief Title: A Low-Carbohydrate Diabetes Prevention Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Kidney Foundation, United States (Other)
Responsible Party: Principal Investigator, Dina Griauzde, Internal Medicine, Clinical Lecturer, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: F046400
Record Dates: First submitted 2017-08-15; First posted 2017-08-23 (Actual); Last update posted 2018-12-12 (Actual); Status verified 2018-12

CONDITIONS: PreDiabetes
MeSH Terms: conditions — Prediabetic State

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Low-Carbohydrate Diabetes Prevention Program (Experimental): At least 20 individuals with prediabetes will participate in a year-long , group-based program.
  Interventions: Behavioral: Low-Carbohydrate Diabetes Prevention Program

INTERVENTIONS:
Behavioral: Low-Carbohydrate Diabetes Prevention Program — LC-DPP participants will be instructed to follow ad-libitum very low-carbohydrate, ketogenic diet, which restricts carbohydrate intake (not including fiber) to 20-35 grams per day with the goal of achieving nutritional ketosis. Participants will be encouraged to eat a normal amount of protein (roughly 80-120 grams per day) and to derive the remaining calories from fat. Allowable foods include: meats, fish, poultry, eggs, cheese, seeds, nuts, leafy greens, non-starchy vegetables, and some fruits.

SUMMARY:
The investigators will conduct a single-arm mixed methods pilot study to estimate weight loss as well as the percentage of participants who achieve 5% weight loss in a 16-week, Low-Carbohydrate Diabetes Prevention Program (LC-DPP). Weight loss from the pilot LC-DPP cohort will be compared to weight loss outcomes from previously published DPP studies. The investigators will also evaluate secondary outcomes including change in physical activity, mental health, psychosocial functioning, and hemoglobin A1c over the 6-month study period.

DETAILED DESCRIPTION:
An estimated 86 million US adults are have prediabetes, and, without intervention, many will develop T2DM over time. Fortunately, T2DM can be prevented or delayed through modest lifestyle changes. The landmark Diabetes Prevention Program (DPP) Trial demonstrated a 58 percent reduction in the 3-year incidence of T2DM among individuals with prediabetes who achieved 7 percent body weight loss and engaged in routine physical activity. Accordingly, the DPP lifestyle intervention has been translated to communities across the United States, and, on average, participant weight change is 4 percent at 12 months. Thus, while group-based DPPs and can effectively promote weight loss among some participants, many DPP participants do not achieve the program goal of 5 to 7 percent body weight loss.

Novel strategies to help participants achieve DPP weight-loss goals are important for two key reasons. First, weight loss is the primary driver of T2DM risk reduction, and the potential population health impact of the intervention is diminished when participants do not lose weight. Second, a growing number of health plans including Medicare offer coverage for the DPP and proposed reimbursement is largely tied to weight loss of at least 5 percent at 6 months and 12 months. The DPP costs approximately $400-$500 per participant per year. Unfortunately, organizations that offer the DPP may be reimbursed for much less than this if participants do not meet weight loss goals, which could significantly compromise the program's long-term financial sustainability.

One promising approach to help DPP participants lose more weight may be through a low-carbohydrate (LC) dietary intervention. Consistent with United States Dietary Guidelines (USDG), the original DPP Trial and translational group-based curricula recommend a low-fat (LF), calorie-restricted diet. However, there is growing controversy regarding the scientific merit of the Dietary Guidelines as well as growing recognition that LC diets may be more effective than LF diets for short-term weight loss and long-term weight maintenance. Notably, weight loss occurs without calorie restriction and LC diets improve blood glucose levels among individuals with T2DM and insulin resistance. Thus, a LC dietary intervention for prediabetes may augment individual weight loss and T2DM risk reduction while also maximizing third-party reimbursement.

The aim of this mixed methods pilot study is to test whether a LC-DPP may lead to greater weight loss than the original DPP. In addition to objective measures of this program's preliminary efficacy (e.g. weight, HbA1c) the study team will also obtain qualitative participant feedback on the intervention. Taken together, these data will be used to improve the curriculum and inform a larger-scale intervention.

ELIGIBILITY:
Inclusion criteria:

1. Overweight, defined as BMI≥25 kg/m2 [31]
2. HbA1c between 5.7-6.4% drawn within 6 months of the study start date
3. Willingness to participate in group-based classes
4. Able to engage in at least light physical activities such as walking.

Exclusion criteria:

1. History of type 1 diabetes or type 2 diabetes
2. Current participation in another lifestyle or behavior change program or research study
3. Vegetarian or vegan lifestyle
4. History of bariatric surgery
5. Inability to read, write, or speak English
6. Inability to provide informed consent
7. Women who are pregnant or intend to become pregnant during the intervention period.
8. Insured by Premier Care or Grad Care; these individuals have the opportunity to participate in a standard DPP, which is offered as a covered benefit through their health plan.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2017-09-11 (Actual); Primary Completion 2018-11-07 (Actual); Study Completion 2018-11-07 (Actual)

PRIMARY OUTCOMES:
Change in body weight per participant over the study period | Baseline, 12 months
  Measured as percent body weight loss per participant
Percentage of participants who achieve weight loss goal | Baseline,12 months
  Measured as percentange of participants who achieve 5% total body weight loss

SECONDARY OUTCOMES:
Change in self-reported weekly physical activity minutes | Baseline, 12 months
  Participants will maintain a log of weekly physical activity minutes
Change in physical activity measured using the International Physical Activity Questionnaire | Baseline, 12 months
  Participants will complete this validated survey
Change in food cravings measured using the Control of Eating Questionnaire | Baseline, 12 months
  Participants will complete this validated survey
Change in stress eating measured using the Palatable Eating Motives Scale | Baseline, 12 months
  Participants will complete this validated survey
Change in self-reported health measured using the Global Health PROMIS Questionnaire | Baseline, 12 months
  Participants will complete this validated survey
Change in autonomous motivation measured using the Treatment Self-Regulation Questionnaire | Baseline, 12 months
  Participants will complete this validated survey
Change in hemoglobin A1c | Baseline, 12 months
  Measured using a laboratory blood draw
Session attendance | Baseline, 12 months
  Measured as the number of sessions attended per participant
Study attrition | Baseline, 12 months
  Number of participants lost to follow-up

OTHER OUTCOMES:
Change in diet as assessed by qualitative review of foods logs | Baseline, 12 months
  Participants will maintain weekly food logs
Change in diet as assessed by response to survey questions | Baseline, 12 months
  Participants will respond to exploratory survey questions about diet created by the study team.
Change in physical symptoms | Baseline, 12 months
  Participants will respond to exploratory survey questions about physical symptoms created by the study team.

CONTACTS AND LOCATIONS:
Locations (1):
- Michigan Medicine, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hafez Griauzde D, Saslow L, Patterson K, Ansari T, Liestenfeltz B, Tisack A, Bihn P, Shopinski S, Richardson CR. Mixed methods pilot study of a low-carbohydrate diabetes prevention programme among adults with pre-diabetes in the USA. BMJ Open. 2020 Jan 21;10(1):e033397. doi: 10.1136/bmjopen-2019-033397. PMID 31969366